CLINICAL TRIAL: NCT01120925
Title: Comparison of Therapeutic Outcome of Twice Transplantation of CD133+ and MNC BM Derived Stem Cells in Cirrhotic Patients: Clinical Trial, Double Blind, Phase I/II
Brief Title: Autologous Bone Marrow Derived Stem Cells in Decompensate Cirrhotic Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Collaborators: University of Tehran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Royan-Liver-002
Record Dates: First submitted 2010-05-08; First posted 2010-05-11 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2010-05

CONDITIONS: Liver Cirrhosis
Keywords: Cirrhotic; Stem Cells; Bone marrow stem cells; Decompensate Cirrhotic Patients
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MNC (Experimental): Bone marrow derived MNC
  Interventions: Biological: MNC
- CD133 (Experimental): CD133 derived from Bone marrow
  Interventions: Biological: CD133
- Control (Placebo Comparator): Normal saline with 5% Human Serum Albumin
  Interventions: Biological: Control

INTERVENTIONS:
Biological: MNC — 2-3 X 109 cells in 20ML suspension IPV in 4 min
  Arms: MNC
Biological: CD133 — 5-15 X 106 cells in 20ML suspension IPV
  Arms: CD133
Biological: Control — Injection of 20 ml Normal saline via IPV
  Arms: Control

SUMMARY:
Liver cirrhosis (LC) is the final outcome for chronic liver diseases. The liver transplantation is the sole effective therapy available to these patients. However, limited number of donors, post surgical complications, immunological rejection, and financial consideration are it's crucial problems. The plasticity of stem cells in bone marrow (BM) to differentiate into Hepatocyte cells was recently confirmed, and several clinical studies have applied BMC injection to induce regeneration of myocardium and blood vessels. In this study, the investigators will study safety and feasibility of twice transplantation of Autologous bone derived marrow mono nuclear (BM-MNC) and enriched CD133+ hematopoietic stem cell through the portal vein in patients with decompensate cirrhosis.

DETAILED DESCRIPTION:
BM Aspiration will be done twice (3months interval) from the iliac crest according to standard procedures under general anesthesia and is collected (200ML) in plastic bags containing anti coagulant. After precipitation of red blood cells, mononuclear cells will be collected by centrifugation in Ficoll-Paque density gradient. For separation of CD133+ cells the CliniMACS instrument will be used. Cells are injected twice (3months interval) via portal vein under sonography monitoring. After cell therapy, patients are followed up every week for 6 months, and laboratory data are analyzed for 6 months

ELIGIBILITY:
Inclusion Criteria:

* 16-65 Years cirrhotic patient
* Approved cirrhosis by elastografy ,biopsy, sonography
* Serum ALT 1/5 times more than normal
* MELD score 12 or Child score B or C

Exclusion Criteria:

* Portal vein thrombosis
* Hepatic encephalopathy, score 3&4
* ALT & AST 3times more than normal
* Serum Cr more than 1/5mg/dL
* (Anti-HIV +) (Anti-HCV+) (HBS-Ag+)
* Hepatocel carcinoma
* Primary sclerosing cholangitis (PSC)
* Esophageal varices grade 4
* Addiction

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Liver function test | 6 months
  Meld score, Child score

SECONDARY OUTCOMES:
Cirrhosis Mortality | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Royan Institute; Reza Malekzadeh, MD, Study Chair — Gastroenterology and hepatic disease research center; Hossein Baharvand, PhD, Principal Investigator — Royan Institute; Mohammad Bagheri, MD, Principal Investigator — Gastroenterology and hepatic disease research center; Massoud Vosough, MD, Study Director — Royan Institute; Nasser Aghdami, MD., PhD, Principal Investigator — Royan Institute
Locations (1):
- Gastroenterology and hepatic disease research center, Tehran, Tehran Province, Iran

REFERENCES:
- See also: Related Info — http://www.royaninstitute.org